CLINICAL TRIAL: NCT01071759
Title: Effects of Dietary Heme/Non-heme Iron and Hp Infection on Maternal Iron-deficiency Anemia and Fetal Growth Outcomes - a Perinatal Longitudinal Study
Brief Title: Effects of Dietary Heme/Non-heme Iron and Helicobacter Pylori (Hp) Infection on Maternal Iron-deficiency Anemia and Fetal Growth Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: E-DA Hospital (Other)
Other Study IDs: EDAH-D-97(P)014A; EMRP-097-123 (Other: E-DA Hospital)
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Pregnancy; Helicobacter Pylori Infection; Iron-Deficiency Anemia
Keywords: Pregnancy; anemia; Helicobacter pylori; Hemoglobin; Iron; Ferritin
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pregnancy

SUMMARY:
Iron deficiency is considered one of the main nutritional deficiency disorders despite the apparent availability of a high-quality diet even in developed countries, and Iron deficiency anemia (IDA) is the most common form of anemia in the world. IDA during pregnancy has been associated with adverse health consequences for both the mother and her developing fetus. Helicobacter pylori (Hp) may be the most common bacterial infection worldwide, infecting almost half of people in developed countries and 80% of people in developing countries. The available data on the prevalence of Hp infection in Taiwan population was 54.4%. We all know that infection with Hp is strongly associated with peptic ulcer and gastric cancer, but recent evidence suggests that Hp is associated with iron deficiency and anemia, although the mechanisms remain unclear. Till now, only few previous studies specifically have addressed a potential role of Hp infection on anemia or iron deficiency during pregnancy. Our previous Research showed, between the Hp infection (+) and Hp infection (-) gravidas, the associations between the Hp infection and iron deficiency were stronger, although not statistically significant. This might be due to that we needed more cases and evidences to prove the relationship between maternal Hp infection and serum iron, ferritin and hemoglobin levels, or we should further consider the interactions of the particular customs or diet preference of the Taiwanese gravidas. This longitudinal study will recruit 140 women from the antenatal care clinics of E-Da Hospital to examine the association between Hp infection and maternal IDA. The standardized interviews of mothers (anthropometric data, socioeconomic status, medical history, obstetric history, alcohol consumption during pregnancy, and history and duration of iron supplementation during pregnancy) will be conducted, Hp infection status will be determined by the urea breath test and IgG enzyme immunoassay, and the measurement of hemoglobin, iron, and ferritin levels will be obtained 5 times at various antepartum and postpartum points of time during pregnancy (routine prenatal visits of 1st, 2nd, and 3rd trimester, puerperium and 2 weeks after delivery). We hope that we could investigate the possible role of Hp infection in iron deficiency and iron-deficiency anemia during pregnancy in Taiwan, and that early detection and treatment of anemia may reduce the risk of blood transfusion and perinatal and maternal mortality.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Ladies

Exclusion Criteria:

* Thalassemia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant Ladies
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2009-02

CONTACTS AND LOCATIONS:
Locations (1):
- E-DA Hospital, Kaohsiung County, Taiwan